CLINICAL TRIAL: NCT01274715
Title: Behavioral Health Coaching for Rural Veterans With Diabetes and Depression
Brief Title: HOPE Pilot for Veterans With Complex Diabetes
Acronym: HOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Collaborators: South Central VA Mental Illness Research, Education & Clinical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Aanand Naik, Assistant Professor of Medicine, Michael E. DeBakey VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VA ID 10G09.H
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Results first posted 2014-05-08 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-04

CONDITIONS: Diabetes; Depression
Keywords: Behavioral health coaching; Diabetes; Emotional health
MeSH Terms: conditions — Diabetes Mellitus; Depression; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Behavioral Health Coaching arm (Experimental): This is a single-arm, pilot study of a health behavior coaching intervention to consist of 12 sessions of coaching over a 3 month period. There is no control arm for this pilot study.
  Interventions: Behavioral: Behavioral Health Coaching

INTERVENTIONS:
Behavioral: Behavioral Health Coaching — Behavioral health coaching consisting of goal-setting, action planning, behavioral activation, and cognitive therapy is delivered by telephone over approximately 3 months.

SUMMARY:
The purpose of this study is to determine if behavioral health coaching for rural veterans with diabetes and depression will improve self-management behaviors and lead to improvement in diabetes care outcomes (e.g., HA1C) and improvement in reported depressive symptoms.

DETAILED DESCRIPTION:
The co-occurence of diabetes and depression is highly prevalent and has dramatic consequences for quality of life and health. Due to the complex interrelation between diabetes and depression, patients often experience both psychological and physiological difficulties. These comorbid problems demand focused interventions that blend physical and emotional health treatments with self-management strategies.Rural-dwelling veterans with diabetes and depression are typically treated in community-based outpatient clinics (CBOCs). Patients with diabetes in rural areas tend to have more problems controlling their blood sugar, blood pressure and cholesterol compared to urban patients; thereby increasing their risk of diabetic complications. Similarly, rural patients with depression have similar barriers to care that increase their risk of poorer health outcomes as well. Using behavioral health coaches (BHCs)to deliver telephone-mediated therapies may enhance the reach of treatments for co-occurring diabetes and depression. The implementation of such treatments requires the development and testing of therapeutic manuals and BHC training protocols to ensure standardization and effectiveness. The BHC intervention has been labeled Health Outcomes through Patient Empowerment (HOPE) and will be offered to eligible patients receiving care through MEDVAMC and its CBOCs. Preliminary data obtained through this pilot grant is to support a larger VA grant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes and Primary Care Physician intent to treat
* Clinically significant symptoms of depression per self-report
* HA1C average of 7.5 or greater in past 12 months AND no HA1C < 7.0 in past 12 months.

Exclusion Criteria:

* Factors that render a telephone-based behavioral activation intervention inappropriate
* Significant cognitive impairment
* Meet criteria of bipolar, psychotic or substance abuse disorder
* Serious medical issues; e.g., terminal cancer
* Reports severe depression or suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aanand D Naik, MD, Principal Investigator — Michael E. DeBakey VA Medical Center; Jeffrey A Cully, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center
Locations (1):
- MEDVAMC, Houston, Texas, United States

REFERENCES:
- [Result] Naik AD, White CD, Robertson SM, Armento ME, Lawrence B, Stelljes LA, Cully JA. Behavioral health coaching for rural-living older adults with diabetes and depression: an open pilot of the HOPE Study. BMC Geriatr. 2012 Jul 24;12:37. doi: 10.1186/1471-2318-12-37. PMID 22828177

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period lasted from January 2011 through July 2011. After patients were screened, recruitment occurred over the phone, where they gave audio consent to participate in the study.
Pre-assignment Details: Three participants who gave consent to participate in the study met exclusion criteria at baseline and were removed from the study before being assigned to the intervention.
Period: Overall Study
Arm/Group | Behavioral Health Coaching
Started | 12
Screened Out at Baseline | 3
Completed | 8
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — After consent, met exclusion criteria. | 1
Not completed — After consent, met exclusion criteria. | 1
Not completed — After consent, met exclusion criteria. | 1

BASELINE CHARACTERISTICS:
Arm/Group | Behavioral Health Coaching
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (5.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in PHQ-9 (Patient Health Questionnaire-9)Scores
Description: The full name of the measure is the Patient Health Questionnaire-9. This is a self-reported measure of depressive symptoms. This is a nine item measure with a response for each item between 0-3. Total scores on this measure range from 0-27, with 0 being a minimum indicating no depressive symptoms, and 27 being the maximum number and severity of depressive symptoms. The coaching sessions take place over approximately 3 months -- outcomes are measured at baseline, 3 months and again at 6 months. Change from baseline to 3 months was calculated. Then change from baseline to 6 months was calculated.
Time Frame: Baseline, 3 months, and 6 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Behavioral Health Coaching
Number analyzed (Participants) | 8
scores on a scale
  Change from baseline to 3-month, M (SD) | 5.14 (2.27)
  Change from baseline to 6-month, M (SD) | 7.03 (4.43)

2. Primary Outcome: Change in Hemoglobin A1C
Description: Value of Hemoglobin A1C reduction post-intervention. The coaching sessions take place over approximately 3 months -- outcomes are measured at baseline, 3 months and again at 6 months. Change from baseline to 3 months was calculated. Then change from baseline to 6 months was calculated.
Time Frame: baseline, 3 months, and 6 months
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Behavioral Health Coaching
Number analyzed (Participants) | 8
percentage of glycated hemoglobin
  Change from baseline to 3 months | 1.13 (1.7)
  Change from baseline to 6 months | 0.84 (1.62)

ADVERSE EVENTS:
Arm/Group | Behavioral Health Coaching
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
A very small sample was collected, and there was not a control group to compare to our intervention group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes